CLINICAL TRIAL: NCT00625209
Title: Phase III of Recombinant Human Activated Protein C and Low Dose of Hydrocortisone and Fludrocortisone in Adult Septic Shock
Brief Title: Activated Protein C and Corticosteroids for Human Septic Shock
Acronym: APROCCHS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Versailles (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); Ministry of Health, France (Other Government)
Responsible Party: Principal Investigator, Djillali Annane, Professor in medicine, University of Versailles
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P070128
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Septic Shock
Keywords: septic shock; coagulation; immunomodulation; survival
MeSH Terms: conditions — Shock, Septic; Thrombosis | interventions — Hydrocortisone; Fludrocortisone; drotrecogin alfa activated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): placebo of hydrocortisone, placebo of fludrocortisone and placebo of activated protein C
  Interventions: Drug: placebos
- 2 (Active Comparator): Hydrocortisone plus fludrocortisone and a placebo of activated protein C
  Interventions: Drug: hydrocortisone and fludrocortisone and placebo
- 3 (Active Comparator): placebo of hydrocortisone, placebo of fludrocortisone and activated protein C
  Interventions: Drug: recombinant human activated protein C and placebos
- 4 (Active Comparator): hydrocortisone plus fludrocortisone plus activated protein C
  Interventions: Drug: recombinant human activated protein C and hydrocortisone and fludrocortisone

INTERVENTIONS:
Drug: placebos — placebo of hydrocortisone as an iv bolus every 6 hours for seven days plus placebo of fludrocortisone given through the nasogastric tube once a day for seven days plus placebo of activated protein C given as a continuous infusion for 96 hours
  Arms: 1
Drug: hydrocortisone and fludrocortisone and placebo — hydrocortisone will be given as 50mg iv bolus every 6 hours for seven days and a tablet of 50µg of fludrocortisone will be given once a day via the nasogastric tube for seven days and a placebo of activated protein C will be given as a continuous infusion for 96 hours
  Arms: 2
Drug: recombinant human activated protein C and placebos — activated protein C will be given as a continuous infusion at a dose of 24 µg/kg/h four 96 hours and hydrocortisone placebo as an iv bolus every 6 hours and fludrocortisone placebo once a day through the gastric tube will be given for seven days
  Arms: 3
Drug: recombinant human activated protein C and hydrocortisone and fludrocortisone — 96 hours continuous infusion of 24µg/kg/h of activated protein C plus seven day treatment with 50mg iv bolus of hydrocortisone every 6 hours and 50µg of fludrocortisone via the nasogastric tube once a day
  Arms: 4

SUMMARY:
This study aims at comparing the efficacy and safety of recombinant human activated protein C to that of low dose of corticosteroids and at investigating the interaction between these drugs in the management of septic shock

DETAILED DESCRIPTION:
Septic shock still places a burden in the healthcare system round around the world. In the early 20ties, clinical trials suggested potential benefits from activated protein C in severe sepsis and of corticosteroids when given to adults with refractory shock. More recent studies suggested that patients with moderate sepsis or septic shock may not benefit from either activated protein C or corticosteroids. Therefore, current international guidelines suggest that physicians may consider using these drugs in the more severe cases of sepsis. The main risk associated with the use of activated protein C is bleeding and the main risk associated with the use of steroids is superinfection. It is paramount that a new adequately powered trial explores the benefit/risk ratio of these two drugs and of their combination in a population of adult patients with septic shock.

After the withdrawal of Xigris in October 2011, the study was suspended and restarted in June 2012 to investigate the benefit to risk ratio of corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized in intensive care unit for less than 7 days
* septic shock for less than 24 hours
* at least one proven site of infection
* at least 2 organ dysfunction as defined by a SOFA score =or> to 3 for at least 6 consecutive hours
* need for vasopressor (dopamine =or>15µg/kg/min or epinephrine/norepinephrine at =or>0,25 µg/kg/min for at least 6 consecutive hours, to maintain systolic arterial pressure at 90 mmHg or more OR mean arterial pressure at 6( mmHg or more
* informed consent

Exclusion Criteria:

* pregnancy or breath feeding
* decision not to resuscitate
* underlying disease with an estimated life expectancy of less than 1 month
* formal indication for corticosteroids
* recent surgery (ie within the past 72 hours) or a surgery at high risk of bleeding
* gastro-intestinal bleeding within the past 6 weeks
* chronic liver disease (Child C)
* recent trauma (ie within the past 72 hours)
* intracranial process
* history of stroke, CNS bleeding or traumatic brain injury within the past 3 months
* platelet counts of less than 30000 per cubic millimeter
* formal indication for curative anticoagulant; prophylactic use of heparin is allowed
* any condition of high risk of bleeding as per patient's primary physicians
* hypersensitivity of activated drotrecogin alpha or any other component of the drug
* no affiliation to a social security

Amendments to eligibility criteria were:

On 27/03/2008: Changes in following exclusion criteria :

* "surgical procedure in the past 7 days" was changed for "surgical procedure within 72 hours, or any surgery associated with high risk of bleeding, or a planned surgery within 24 h".
* "chronic liver disease" was clarified as "chronic liver disease with Child score C".
* "severe thrombopenia" was clarified "as severe thrombopenia (<30,000/mm3, before transfusion).

On 25/08/2009: The exclusion criteria: surgical procedure within 72 hours, or any surgery associated with high risk of bleeding, or a planned surgery within 24 h" was changed for "surgical procedure within 12 hours, or any surgery associated with high risk of bleeding

On 11/06/2010: the inclusion criteria: admitted to the ICU for < 7 days was removed; and a new exclusion criteria was added: "patients who had a previous episode of sepsis during the same hospital stay

On 18/04/2012: following the withdrawal of DAA from the market: the following exclusion criteria (only related to DAA) were removed :

1. any surgery in the past 12 hours, or any surgery associated with high risk of bleeding;
2. chronic liver disease with a Child score C;
3. recent trauma;
4. any intracranial mass, or stroke or head injury in the past 3 months;
5. severe thrombocytopenia (< 30.000 /mm3, before platelet transfusion);
6. formal indication for anticoagulation, or any other condition associated with increased risk of bleeding, as appreciated by the patient's physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1241 (Actual)
Dates: Start 2008-03; Primary Completion 2015-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
90-day mortality | 90 day

SECONDARY OUTCOMES:
mortality at 28 day | 28-day
mortality at ICU discharge | ICU discharge
mortality at hospital discharge | hospital discharge
mortality at 6 months | 6 months
decision to withhold or withdraw active treatments | up to 90 days
Time to wean vasopressor therapy | up to 90 days
number of days alive and free of vasopressor therapy | up to 90 days
time to achieve an SOFA score of less than 6 | up to 90 days
number of days alive with a SOFA score < 6 points | up to 90 days
time to wean mechanical ventilation | up to 90 days
number of days alive and free of mechanical ventilation | up to 90 days
Length of intensive care unit and hospital stay | up to hospital discharge
acquisition of new infection | up to 180 days
new episode of sepsis | up to 90 days
new episode of septic shock | up to 90 days
bleeding events | up to 90 days
neurological sequels at intensive care unit and at hospital discharge and at 90 and 180 days | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Misset, MD, Principal Investigator — Unity Health Toronto; Claude Martin, MD, Principal Investigator — Assistance Publique Hopitaux de Marseille, hôpital Nord; Alain Cariou, MD, Principal Investigator — Assistance Publique Hôpitaux de Paris, Hôpital Cochin; Jean Carlet, MD, Principal Investigator — Unity Health Toronto; Christian Brun Buisson, MD, Principal Investigator — Assistance Publique Hôpitaux de Paris, Hôpital Henri Mondor; Djillali Annane, MD, Principal Investigator — Assistance Publique Hôpitaux de Paris, Hôpital Raymond Poincaré
Locations (4):
- France (4):
  - Henri Mondor Hospital, Créteil
  - Raymond Poincaré Hospital, Garches
  - Pitié Salpêtrière Hospital, Paris
  - Saint Josef Hospital, Paris

REFERENCES:
- [Background] Annane D, Buisson CB, Cariou A, Martin C, Misset B, Renault A, Lehmann B, Millul V, Maxime V, Bellissant E; APROCCHSS Investigators for the TRIGGERSEP Network. Design and conduct of the activated protein C and corticosteroids for human septic shock (APROCCHSS) trial. Ann Intensive Care. 2016 Dec;6(1):43. doi: 10.1186/s13613-016-0147-3. Epub 2016 May 6. PMID 27154719
- [Result] Annane D, Timsit JF, Megarbane B, Martin C, Misset B, Mourvillier B, Siami S, Chagnon JL, Constantin JM, Petitpas F, Souweine B, Amathieu R, Forceville X, Charpentier C, Tesniere A, Chastre J, Bohe J, Colin G, Cariou A, Renault A, Brun-Buisson C, Bellissant E; APROCCHSS Trial Investigators. Recombinant human activated protein C for adults with septic shock: a randomized controlled trial. Am J Respir Crit Care Med. 2013 May 15;187(10):1091-7. doi: 10.1164/rccm.201211-2020OC. PMID 23525934
- [Derived] Heming N, Renault A, Kuperminc E, Brun-Buisson C, Megarbane B, Quenot JP, Siami S, Cariou A, Forceville X, Schwebel C, Leone M, Timsit JF, Misset B, Benali MA, Colin G, Souweine B, Asehnoune K, Mercier E, Chimot L, Charpentier C, Francois B, Boulain T, Petitpas F, Constantin JM, Dhonneur G, Baudin F, Combes A, Bohe J, Loriferne JF, Cook F, Slama M, Leroy O, Capellier G, Dargent A, Hissem T, Bounab R, Maxime V, Moine P, Bellissant E, Annane D; APROCCHSS investigators; CRICS-TRIGGERSEP network. Hydrocortisone plus fludrocortisone for community acquired pneumonia-related septic shock: a subgroup analysis of the APROCCHSS phase 3 randomised trial. Lancet Respir Med. 2024 May;12(5):366-374. doi: 10.1016/S2213-2600(23)00430-7. Epub 2024 Feb 1. PMID 38310918
- [Derived] Annane D, Renault A, Brun-Buisson C, Megarbane B, Quenot JP, Siami S, Cariou A, Forceville X, Schwebel C, Martin C, Timsit JF, Misset B, Ali Benali M, Colin G, Souweine B, Asehnoune K, Mercier E, Chimot L, Charpentier C, Francois B, Boulain T, Petitpas F, Constantin JM, Dhonneur G, Baudin F, Combes A, Bohe J, Loriferne JF, Amathieu R, Cook F, Slama M, Leroy O, Capellier G, Dargent A, Hissem T, Maxime V, Bellissant E; CRICS-TRIGGERSEP Network. Hydrocortisone plus Fludrocortisone for Adults with Septic Shock. N Engl J Med. 2018 Mar 1;378(9):809-818. doi: 10.1056/NEJMoa1705716. PMID 29490185